CLINICAL TRIAL: NCT04843410
Title: Effect of Exercise in the Management of Chemotherapy-Related Peripheral Neuropathy
Brief Title: Effect of Exercise in the Management of Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Necmiye Comlekci, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 13022260-300-180785
Record Dates: First submitted 2021-04-10; First posted 2021-04-13 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; Chemotherapeutic Toxicity
Keywords: peripheral neuropathy, chemotherapy, exercise, oncology
MeSH Terms: conditions — Peripheral Nervous System Diseases; Motor Activity; Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Exercise group (Experimental): In this prospective study, patients who applied to Zonguldak Atatürk State Hospital Oncology Outpatient Clinic received at least three cures of taxane and platinum-based treatment (monotherapy or combined) and developed grade 2 and higher peripheral neuropathy (lung cancer, breast cancer) as a result of motor and sensory neuropathy evaluation. , gynecological cancers, colorectal cancers), patients with stable vital signs who can tolerate the exercise, patients without bone metastases, patients older than 18 years of age, and patients who agree to participate in the study.
  The experimental group will be taught an exercise program to apply regularly twice a day. The researcher will give the patient the barbed ball and barbed roller required for the exercise. In addition, visual training material will be given for the exercise program so that the patient can repeat the training whenever he wants to ensure the permanence of the patient education.
  Interventions: Other: Hand-foot exercise
- The routine care: Control Group (Sham Comparator): In this prospective study, patients who applied to Zonguldak Atatürk State Hospital Oncology Outpatient Clinic received at least 3 cures of taxane and platinum-based treatment (monotherapy or combined) and developed grade 2 and higher peripheral neuropathy (lung cancer, breast cancer) as a result of motor and sensory neuropathy evaluation. , gynecological cancers, colorectal cancers), patients with stable vital signs, patients without bone metastases, patients older than 18 years of age, and patients who agree to participate in the study. The routine care of the clinic will be applied to the control group.
  Interventions: Other: The routine care

INTERVENTIONS:
Other: Hand-foot exercise — The experimental group will be taught a regular exercise program for 15 minutes twice a day. The sensory exercise ball required for exercise will be given to the patients by the researcher. In addition, visual training material will be provided for the exercise program so that the patient can repeat the training at any time to ensure the permanence of the patient education. The standard care protocol of the clinic will be applied to the control group.
  Arms: Experimental: Exercise group
Other: The routine care — Education about chemotherapy-associated peripheral neuropathy risk factors, why it develops and its management
  Arms: The routine care: Control Group

SUMMARY:
Chemotherapy-associated peripheral neuropathy is a common complication in patients receiving taxane and platinum-based chemotherapy. Peripheral neuropathy may cause the patient's daily life activities to be hindered, quality of life to deteriorate, treatment dose reduced, or even discontinuation of treatment. In the literature, different studies have been carried out using many pharmacological and non-pharmacological approaches in the management of this problem, but so far, any approach that has been shown to be effective in its management has not been clearly defined. One of the approaches whose effectiveness is evaluated in management is exercise. There have been published case reports and several experimental studies examining small patient groups on this subject, and it has been shown to have significant benefits in the management of peripheral neuropathy. This study was planned to determine whether exercise is an effective method in the management of chemotherapy-associated peripheral neuropathy in oncology patients.

DETAILED DESCRIPTION:
Chemotherapy-associated peripheral neuropathy is a common complication in patients undergoing taxane and platinum-based chemotherapy. Peripheral neuropathy may cause the patient's activities of daily living to be inhibited, deterioration of quality of life, reduction of treatment dose, and even discontinuation of treatment. In the literature, different studies have been carried out using many pharmacological and non-pharmacological approaches to manage this problem, but no approach that has been shown to be effective in its management has not been clearly defined until now. One of the approaches whose effectiveness is evaluated in management is exercise. Published case reports and a few experimental studies examining small patient groups have been found to have significant benefits in the management of peripheral neuropathy. This study was planned to determine whether exercise is effective in managing associated peripheral neuropathy in oncology patients.

General Information Cancer is one of the most important health problems in the world and our country. Despite significant developments in cancer treatment, treatment-related side effects can lead to adverse effects on the quality of life of patients, limitation of their activities, and even restriction of the treatment dose and discontinuation of the treatment, which may adversely affect the response of the patient to treatment.

Antineoplastic agents used in cancer treatment provide treatment of cancer or prevent its progression by preventing the division and proliferation of cancer cells. However, these drugs cause many important side effects such as anemia, diarrhea, nausea, vomiting, infections, fatigue, alopecia, infertility, pain, and peripheral neuropathy in the patient by affecting not only cancer cells but also normal cells and body structures.

Peripheral neuropathy is a significant side effect that adversely affects patients' quality of life receiving taxane or platinum-based chemotherapy. The incidence of chemotherapy-associated peripheral neuropathy varies between 19 and 85%, depending on the type of chemotherapy protocol administered, the drug dose used in the treatment, and the duration of administration. The incidence of peripheral neuropathy, according to the type of antineoplastic agent applied, is between 70-100% in platinum-administered patients, 11-87% in taxane-administered patients, 20-60% in thalidomide-administered patients, and 60-65% in ixabepilone-administered patients. The most common antineoplastic agents causing peripheral neuropathy are platinum (oxaliplatin and cisplatin), vinca alkaloids (vincristine and vinblastine), and taxanes (paclitaxel, docetaxel), proteasome inhibitors (bortezomib), and immunomodulatory drugs (thalidomide). These chemotherapeutic agents, which cross the blood-brain barrier, affect the dorsal root ganglia and peripheral axons in the spinal cord, causing changes in motor, sensory and autonomic neurons, causing the development of peripheral neuropathy.

Many factors such as age, concomitant diabetes mellitus history, microtubules or mitochondrial damage, oxidative stress, changes in ion channel activity, and damage to the myelin sheath play a role in the development of peripheral neuropathy. Sensory, motor, and autonomic symptoms may develop in patients with chemotherapy-related peripheral neuropathy. First, patients develop sensory symptoms such as numbness in the hands and feet, tingling, change in the sense of touch, paresthesia, dysesthesia, and patients usually describe these sensory changes as a feeling of wearing gloves and socks. As the picture progresses, spontaneous burning, fever, electric shock, mechanical or thermal allodynia, and hyperalgesia may also develop in patients. In severe cases, these symptoms can go as far as loss of sensory perception. Muscle weakness, gait, and balance disorders that increase the risk of falling are frequently reported motor symptoms by patients. Orthostatic hypotension, constipation, urinary dysfunction, and sexual dysfunction are common autonomic symptoms in patients. While these symptoms improve over time with the discontinuation of chemotherapy in some patients, they can be permanent because neuron damage occurs in most patients. Therefore, approaches presented in the management of peripheral neuropathy in the literature are quite limited.

In a systematic review of the effectiveness of pharmacological approaches in the management of chemotherapy-associated peripheral neuropathy, it was reported that the use of pharmacological agents such as duloxetine, gabapentin, acetyl-L-carnitine (ALC), amitriptyline, cannabinoid, lamotrigine, and topical baclofen could be recommended in the management of this problem. However, studies evaluating the efficacy of these pharmacological agents were found to be insufficient in terms of evidence.

Non-pharmacological approaches whose effectiveness has been evaluated in the management of chemotherapy-related peripheral neuropathy are acupuncture, acupressure, neurofeedback, scrambler therapy, cold application, reflexology, massage, exercise, relaxation techniques, physical therapy, and magnetic therapy.

Exercise, one of these approaches, has been reported to be effective in reducing pain, numbness, tingling, loss of sensation, and increasing muscle strength and balance due to peripheral neuropathy in different patient groups. In a quasi-experimental study conducted on patients with a modified neuropathy score (range 0-20) of 5 and above, it was observed that closed kinetic exercises decreased the neuropathy score and increased the balance. A 10-week home-based exercise program for breast cancer patients has been shown to improve symptoms of peripheral neuropathy. In a randomized controlled study with patients with metastatic colorectal cancer, resistance and balance exercises were applied to the experimental group for eight weeks. According to the results of the study, when the experimental group and the control group were compared, peripheral neuropathy symptoms remained the same, while a significant improvement was found in balance functions. In the study of Bland et al., it was stated that exercise significantly improved the CIPN20 score and reduced peripheral neuropathy in patients with breast cancer receiving taxane therapy. However, although the number of studies showing exercise efficacy in managing chemotherapy-associated peripheral neuropathy is quite limited, studies with small samples have low evidence strength.

This study was planned to determine whether exercise is an effective approach in the management of chemotherapy-associated peripheral neuropathy in oncology patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received at least 3 cycles of taxane and platinum-based treatment (monotherapy or combined) and developed grade 2 or higher peripheral neuropathy as a result of motor and sensory neuropathy evaluation (lung cancer, breast cancer, gynecological cancers, colorectal cancers), Patients with stable vital signs who can tolerate exercise,
* No bone metastases,
* Patients older than 18 years old,
* Patients who agree to participate in the study will participate.

Exclusion Criteria:

* Newly starting chemotherapy, Peripheral neuropathy due to problems other than chemotherapy (tumor compression, nutritional disorders, infections and systemic diseases such as diabetes mellitus), Vital signs that cannot tolerate exercise are non-stable, Bone metastases,
* Patients with impaired skin integrity in their hands and feet and who do not agree to participate in the study will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Patient Information Form | Baseline (first meeting (start the study))
  Patient Information Form: The patient information form developed by the researcher in line with the literature will be used in collecting data. The patient information form consists of 5 sections: personal characteristics, economic status, information about the health process, information about peripheral neuropathy and information about the disease process.
Common Terminology Criteria for Adverse Events (CTCAE) - Version 5.0 Classification | 8 weeks
  Common Terminology Criteria for Adverse Events (CTCAE) - Version 5.0 Classification: The CTCAE 5.0 classification was designed by the American National Cancer Institute (NCI) to broadly describe and rank adverse reactions that may arise from a variety of causes. A rating (severity) scale is given for each side effect term. In this classification, grad indicates the severity of the side effect. The severity of adverse events were graded: grade 1 (mild), grade 2 (moderate), grade 3 (severe), grade 4 (life threatening), and grade 5 (side effect-related death).
European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | 8 weeks
  The overall quality of life of patients will be assessed using the European Organization for Cancer Research and Treatment Quality of Life Scale. The scale was developed by EORTC, content validity and reliability study was performed by Beşer and Öz in our country, and the Cronbach alpha reliability coefficient was found to be r = 0.9014. The EORTC QLQC30 Version 3.0 quality of life scale is a widely used quality of life assessment tool for patients with cancer. The EORTC-QLQ-C30 consists of 30 questions and three subtitles: general well-being, functional difficulties and symptom control.
European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Chemotherapy-Induced Peripheral Neuropathy (EORTC QLQ-CIPN20) | 8 weeks
  The EORTC QLQ-CIPN20 is a 20-item assessment tool used to reveal the symptoms of peripheral neuropathy associated with chemotherapy and the effect of functional limitations caused by this problem on patients' lives. Scale to be sensory (tingling, numbness, pain, instability while walking or standing, discriminating temperature and hearing), motor (cramps, writing, grasping small objects, weakness) and autonomic (dizziness after changing position, vision, erectile dysfunction) It has 3 subscales. The 20 items in the scale are Likert-type and the answers are evaluated by giving None "1", a little "2", Rather "3", and a lot of "4" points. High scores from these sections indicate more symptoms and problems, and low scores indicate less symptoms and problems.

CONTACTS AND LOCATIONS:
Overall Officials: Necmiye ÇÖMLEKÇİ, MSc, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
When the research is completed and published, the research data will be shared in the supplementary document.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: For 10 years